CLINICAL TRIAL: NCT03915028
Title: Thermal Cures in the Treatment of Multiple Sclerosis: Effectiveness on the Quality of Life
Brief Title: Thermal Cures in the Treatment of Multiple Sclerosis
Acronym: SPA-SEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A02411-54
Record Dates: First submitted 2019-03-12; First posted 2019-04-16 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Spa treatment; Crenotherapy; Balneotherapy; Physical exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated group by thermal cure (Experimental): Treated group will benefit, within 6 weeks of the inclusion, from the thermal cure in one of the thermal establishments.
  Interventions: Other: Spa therapy
- Control group (No Intervention): Control group will receive a thermal cure after the end of the study

INTERVENTIONS:
Other: Spa therapy — The standardized treatment will consist of 4 spa treatments per day for 3 consecutive weeks.
  Each day, the patient receives at least four treatments, among which:
  * Cure of Drink (in addition to 4 daily cares)
  * Bath in running water: Bath
  * Bath in running water: Pool at 32 ° C
  * Bath with aerobain
  * Immersion shower bath
  * Shower of high pressure under immersion in swimming pool
  * General penetrating shower
  * General jet shower
  * Local jet shower
  * Local mud bath at the feet
  * Single poultice
  * Multiple poultice
  * Compress
  * Mobilization pool
  * Massages under water
  Arms: Treated group by thermal cure

SUMMARY:
Multiple Sclerosis (MS) is a chronic, progressive disease with a high prevalence in France, with significant public health consequences. The benefit of spa treatments on the quality of life in this population has not been evaluated. The methods of study in clinical pharmacology can be a scientific methodological model for the evaluation of thermal practices and it is in this perspective that investigators want to lead this project.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, progressive disease with a high prevalence in France, and its consequences in terms of public health are important. In this disease, the alteration of the quality of life (QoL) is constant and multifactorial : pain, fatigue, decrease in functional capacities, sleep disorders, cognitive disorders, vesico-sphincterian disorders, anomolytic disorders. -rectal and genito-sexual. The benefit of thermal cures on the quality of life in this population has not been evaluated, even if there is some literature in the literature suggesting a benefit of hydrotherapy on equilibrium or on pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient with primary or progressive secondary-phase MS
* Showing EDSS <7 severity criteria
* Patient with MS for whom an indication of spa treatment has been made,
* Patient agreeing to participate in this study and therefore accepting the constraints related to the design "immediate cure-deferred cure",
* Patient receiving the general social security scheme,
* Patient having given written consent to participate in the study

Exclusion Criteria:

* Patient does not meet the inclusion criteria,
* Patient with relapsing remitting MS
* Patient unfit according to the investigator to complete the rating scales
* Patient with heat intolerance called "Uhthoff effect"
* Patient with a contraindication to the spa treatment: urinary or faecal leakage, wound, thrombophlebitis less than three months old, unstabilized cardio respiratory disease.
* Patient with serious life-threatening condition (ie, cancer)
* Patient under tutorship or curatorship
* Patient participating in another interventional clinical research project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Benefit of spa treatment on quality of life assessed by the scale SEP-59 | within 15 weeks after inclusion
  Difference of the score of quality of live assessed by the scale SEP-59 between the patient will receive the immediat spa therapy and the second group which won't receive the spa therapy immediately. SEP-59 is built on the basis of a generic scale, the SF-36. The analysis of SEP-59 is done by computer processing in order to calculate the score of the various axes (pain, physical activity, general wellbeing ...) which are independent (there is no overall score).

SECONDARY OUTCOMES:
Benefit of a spa treatment based on average number of steps per day for one week assessed by actimeter | 9 weeks after inclusion
  Difference of the average number of steps per day for one week between the patient will receive the immediat spa therapy and the second group which won't receive the spa therapy immediately.
Benefit of a thermal cure based on treatment consumption of hospital and ambulatory care | 15 to 17 weeks after inclusion
  Difference of the number of treatment consumption of hospital and ambulatory care between the patient will receive the immediat spa therapy and the second group which won't receive the spa therapy immediately
Benefit of a thermal cure based on depression and anxiety assessed by the scale Hospital Anxiety and depression scale | 15 to 17 weeks after inclusion
  Difference of the level of pain assessed by the scale Hospital Anxiety and depression between the patient will receive the immediat spa therapy and the second group which won't receive the spa therapy immediately.HADS is a self-administered scale of 14 items, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). It contains no somatic item that can be confused with symptomatic manifestations of a disease.
  Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales and for the entire HADS (HADS-T).
  Limit scores distinguish between: non-cases or asymptomatic cases (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11).
Benefit of a thermal cure based on tiredness assesed by the fatigue impact scale | 15 to 17 weeks after inclusion
  Difference of the level of pain assessed by the fatigue impact scale between the patient will receive the immediat spa therapy and the second group which won't receive the spa therapy immediately. It is a self-assessment tool in which the patient is asked to note the extent to which fatigue has caused them problems in certain situations. (0 = no problem, 4 = extreme problems). A maximum score of 160 is obtained for the 40 items.
Benefit of a thermal cure regarding pain assessed by the scale DN 4 | 15 to 17 weeks after inclusion
  Difference of the level of pain assessed by the DN4 scale between the patient will receive the immediat spa therapy and the second group which won't receive the spa therapy immediately

CONTACTS AND LOCATIONS:
Locations (1):
- Département de Médecine Physique et de Réadaptation, Hopital LAPEYRONIE, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided